CLINICAL TRIAL: NCT00195624
Title: A Pilot Study of Alemtuzumab (Campath) in Patients With Relapsed or Refractory Severe Aplastic Anemia
Brief Title: Alemtuzumab to Treat Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050242; 05-H-0242
Record Dates: First submitted 2005-09-16; First posted 2005-09-19 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2018-10

CONDITIONS: Severe Aplastic Anemia, Refractory; Severe Aplastic Anemia, Relapse
Keywords: Immunosuppression; T-cells; Hematopoiesis; Autoimmunity; Thrombocytopenia; Severe Aplastic Anemia; SAA
MeSH Terms: conditions — Anemia, Aplastic; Recurrence; Autoimmune Diseases; Thrombocytopenia | interventions — Alemtuzumab; Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Relapsed severe aplastic anemia (Experimental): Subjects diagnosed with relapsed severe aplastic anemia
  Interventions: Biological: Alemtuzumab (Campath )
- Refractory severe asplastic anemia (Experimental): Subjects diagnosed with refractory severe aplastic anemia
  Interventions: Biological: Alemtuzumab (Campath )
- Relapse after Alemtuzumab (Experimental): Subjects who relapse after initial response to alemtuzumab therapy will have cyclosporine added to the regimen after the 6 month visit.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Biological: Alemtuzumab (Campath ) — Campath administered at a dose of 10/mg/day for 10 days
  Arms: Refractory severe asplastic anemia; Relapsed severe aplastic anemia
Drug: Cyclosporine — Subjects who relapse after initial response to alemtuzumab therapy will have cyclosporine added to the regimen after the 6 month visit. Dosing will be based on ideal body weight and will be adjusted to maintain a target level of 200 - 400 ng /ml.
  Arms: Relapse after Alemtuzumab

SUMMARY:
This study will evaluate the safety and usefulness of a new immunosuppressive drug, alemtuzumab (Campath ), in patients with severe aplastic anemia (SAA). SAA is a rare and serious blood disorder in which the bone marrow stops making red blood cells, white blood cells and platelets. Alemtuzumab is a monoclonal antibody that attaches to and kills white blood cells called lymphocytes. In certain types of aplastic anemia, lymphocytes are responsible for the destruction of stem cells in the bone marrow, leading to a decrease in blood counts. Because alemtuzumab destroys lymphocytes, it may be effective in treating aplastic anemia. Alemtuzumab is currently approved to treat chronic lymphocytic leukemia and is also helpful in other conditions that require immunosuppression, such as rheumatoid arthritis and immune cytopenias.

Patients 2 years of age and older with severe aplastic anemia whose disease does not respond to immunosuppressive therapy or has recurred following immunosuppressive therapy may be eligible for this study. Participants undergo the following tests and procedures:

* Pretreatment evaluation: Patients have a medical history, physical examination, blood tests, electrocardiogram (EKG), echocardiogram, 24-hour Holter monitor (continuous 24-hour monitoring of electrical activity of the heart), bone marrow biopsy (withdrawal through a needle of a small sample of bone marrow for analysis).
* Placement of a central line, if needed: An intravenous line (tube) is placed into a major vein in the patient's chest. It can stay in the body for the entire treatment period and be used to give chemotherapy or other medications, including antibiotics and blood transfusions, if needed, and to withdraw blood samples.
* Alemtuzumab therapy: Patients are admitted to the NIH Clinical Center for the first few injections for close monitoring of side effects. After receiving an initial small test dose, patients begin the first of ten daily injections under the skin, each lasting about 2 hours. Once patients tolerate the infusions with minimal or no side effects, they may be given the remaining infusions on an outpatient basis. Patients who relapse after their initial response to alemtuzumab are given cyclosporine to see if this drug will boost their immune response.
* Patients receive transfusions, growth factors, and antibiotic therapy, as needed.
* Infection therapy: Patients are given aerosolized pentamidine to protect against lung infections and valacyclovir to protect against herpes infections.
* A blood test is done and vital signs are measured every day while patients receive alemtuzumab.
* Patients have an echocardiogram and 24-hour Holter monitor after the last dose of alemtuzumab.
* Blood tests are done weekly for the first 3 months after alemtuzumab administration, then every other week until 6 months.

Patients return to the NIH for follow-up visits 1 month, 3 months, 6 months, and yearly for 5 years after the last dose of alemtuzumab for the following tests and evaluations:

* Blood test
* Repeat echocardiogram at 3-month visit
* Repeat bone marrow biopsy 6 months and 12 months after alemtuzumab, then as clinically indicated for 5 years.

DETAILED DESCRIPTION:
Hematopoietic stem cell destruction in many human bone marrow failure syndromes is now recognized to be secondary to immune mechanisms. Severe aplastic anemia (SAA) is a life-threatening blood disease which can be effectively treated with immunosuppressive drug regimens. However, a significant minority of patients with SAA fail to respond to a single course of horse antithymocyte globulin and cyclosporine, and other patients experience relapse, especially on discontinuation of therapy. Pancytopenia secondary to refractory or relapsed aplastic anemia has a poor prognosis, with death usually resulting from infectious complications. Alemtuzumab (Campath ) is a humanized IgG1 monoclonal antibody directed against the CD52 protein; CD52 is expressed on all lymphocytes and monocytes. Alemtuzumab (Campath ) produces profound and persistent lymphopenia. The antibody has been used to treat a wide range of autoimmune diseases, lymphoid malignancies, and in solid organ and hematopoietic stem cell transplantation. In our limited experience with alemtuzumab for the treatment of SAA refractory to horse antithymocyte globulin, meaningful hematologic responses have been observed and toxicity has been modest.

We therefore propose a non-randomized pilot phase II study of this humanized monoclonal antibody in SAA relapsed or refractory to ATG. Commercially available alemtuzumab (Campath ) will be administered at 10 mg per day subcutaneously for 10 days total.

The primary end point of the study is the response rate at 6 months, defined as no longer satisfying blood count criteria for SAA.

Relapse, robustness of the hematopoietic recovery at 3 and 6 months, 3 months responses, survival, and clonal evolution to myelodysplasia and acute leukemia will be secondary end points.

ELIGIBILITY:
* INCLUSION CRITERIA:

Relapsed severe aplastic anemia after initial hematologic response to a prior course of h-ATG or r-ATG based immunosuppression

Or

Refractory severe aplastic anemia not responding to both horse-ATG and rabbit ATG-based immunosuppression

The criteria for severe aplastic anemia are two of the three criteria:

* Absolute neutrophil count less than or equal to 500 /mm(3)
* Platelets to less than or equal to 20,000/mm(3)
* Absolute reticulocyte count less than 60,000 /microL

Age greater than or equal to 2 years old and greater than 12 kg

Prospective subjects or their parent(s)/responsible guardian(s) must be able to comprehend and be willing to sign an informed consent.

EXCLUSION CRITERIA:

Known Diagnosis of Fanconi's anemia

Evidence of a clonal disorder on cytogenetics. In the refractory disease setting, prospective subjects with super severe neutropenia (ANC less than 200 /microL) will not be excluded if results of cytogenetics are not available or pending.

Infection not adequately responding to appropriate therapy

HIV positivity

Failure to discontinue the herbal supplements Echinacea purpurea or Usnea barbata (Old Man's Beard) within 2 weeks of enrollment

Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within 7-10 days is likely

Previous hypersensitivity to alemtuzumab or its components

Potential subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible

Current pregnancy, or unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential

Not able to understand the investigational nature of the study or give informed consent

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-09-15; Primary Completion 2014-04-14 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Barrett AJ. The treatment of severe acquired aplastic anemia. Blood. 1995 Jun 15;85(12):3367-77. No abstract available. PMID 7780125
- [Background] Young NS, Maciejewski J. The pathophysiology of acquired aplastic anemia. N Engl J Med. 1997 May 8;336(19):1365-72. doi: 10.1056/NEJM199705083361906. No abstract available. PMID 9134878
- [Background] Zoumbos NC, Gascon P, Djeu JY, Trost SR, Young NS. Circulating activated suppressor T lymphocytes in aplastic anemia. N Engl J Med. 1985 Jan 31;312(5):257-65. doi: 10.1056/NEJM198501313120501. PMID 2981406
- [Derived] Aggarwal N, Manley AL, Shalhoub R, Durrani J, Rios O, Lotter J, Patel BA, Wu CO, Young NS, Groarke EM. Alemtuzumab in relapsed immune severe aplastic anemia: Long-term results of a phase II study. Am J Hematol. 2023 Jun;98(6):932-939. doi: 10.1002/ajh.26924. Epub 2023 Apr 6. PMID 37021397
- [Derived] Zaimoku Y, Patel BA, Adams SD, Shalhoub R, Groarke EM, Lee AAC, Kajigaya S, Feng X, Rios OJ, Eager H, Alemu L, Quinones Raffo D, Wu CO, Flegel WA, Young NS. HLA associations, somatic loss of HLA expression, and clinical outcomes in immune aplastic anemia. Blood. 2021 Dec 30;138(26):2799-2809. doi: 10.1182/blood.2021012895. PMID 34724566
- [Derived] Pang Y, Xiao HW, Zhang H, Liu ZH, Li L, Gao Y, Li HB, Jiang ZJ, Tan H, Lin JR, Du X, Weng JY, Nie DN, Lin DJ, Zhang XZ, Liu QF, Xu DR, Chen HJ, Ge XH, Wang XY, Xiao Y. Allogeneic Bone Marrow-Derived Mesenchymal Stromal Cells Expanded In Vitro for Treatment of Aplastic Anemia: A Multicenter Phase II Trial. Stem Cells Transl Med. 2017 Jul;6(7):1569-1575. doi: 10.1002/sctm.16-0227. Epub 2017 May 15. PMID 28504860
- [Derived] Scheinberg P, Nunez O, Weinstein B, Scheinberg P, Wu CO, Young NS. Activity of alemtuzumab monotherapy in treatment-naive, relapsed, and refractory severe acquired aplastic anemia. Blood. 2012 Jan 12;119(2):345-54. doi: 10.1182/blood-2011-05-352328. Epub 2011 Nov 8. PMID 22067384
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-H-0242.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Refractory: Patients who are refractory to prior courses of horse and rabbit antithymocyte globulin (ATG) based immunosuppresive therapy.
- Relapsed: Patients who have responded and relapsed following a prior course of antithymocyte globulin (ATG) based immunosuppresive therapy.
Period: Overall Study
Arm/Group | Refractory | Relapsed
Started | 5 | 42
Completed | 5 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Refractory | Relapsed | Total
Number analyzed (Participants) | 5 | 42 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 6 | 7
  Between 18 and 65 years | 3 | 27 | 30
  >=65 years | 1 | 9 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 24 | 25
  Male | 4 | 18 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 3 | 35 | 38
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 10 | 10
  White | 2 | 23 | 25
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematological Response at 6 Months
Description: Hematological response is defined as no longer satisfying blood count criteria for Severe Aplastic Anemia. Patients were classified as responders if they met two of the following three criteria: ANC greater than 500/ mm'; platelet count greater than 20,000/mm3; and reticulocyte count greater than 40,000/mm3 (60,000/mm3 after January 1993).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Refractory | Relapsed
Number analyzed (Participants) | 5 | 42
Participants | 0 | 18

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Refractory | Relapsed
All-Cause Mortality (participants affected / at risk) | 5/5 | 13/42
Serious Adverse Events (participants affected / at risk) | 2/5 | 22/42
Other Adverse Events (participants affected / at risk) | 4/5 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Refractory (N=5) | Relapsed (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 15
Cardiac failure (Cardiac disorders) | 1 | 0
Presyncope (Cardiac disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Allergic transfusion reaction (Immune system disorders) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Haemorrhagic ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system inflammation (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Vaginal ulceration (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Refractory (N=5) | Relapsed (N=42)
Ecchymosis (Blood and lymphatic system disorders) | 0 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 14
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Petechiae (Blood and lymphatic system disorders) | 1 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Transfusion reaction (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Chest discomfort (Cardiac disorders) | 0 | 3
Chest pain (Cardiac disorders) | 0 | 3
Dizziness (Cardiac disorders) | 0 | 6
Dyspnoea (Cardiac disorders) | 0 | 6
Dyspnoea exertional (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Hyperglycaemia (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 2
Eye swelling (Eye disorders) | 0 | 1
Scleral haemorrhage (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 2
Visual impairment (Eye disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 5
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 8
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1
Oropharyngeal pain (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 4
Asthenia (General disorders) | 0 | 2
Catheter site pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 15
Cold sweat (General disorders) | 0 | 1
Decreased appetite (General disorders) | 1 | 2
Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 12
Feeling cold (General disorders) | 0 | 2
Flushing (General disorders) | 0 | 1
Hot flush (General disorders) | 0 | 1
Hyperhidrosis (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 4 | 25
Injection site inflammation (General disorders) | 0 | 2
Night sweats (General disorders) | 0 | 2
Pain (General disorders) | 0 | 7
Pallor (General disorders) | 0 | 1
Peripheral coldness (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 16
Allergic sinusitis (Immune system disorders) | 0 | 1
Bronchospasm (Immune system disorders) | 0 | 1
Urticaria (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 6
Urinary tract infection (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 11
Iron overload (Injury, poisoning and procedural complications) | 0 | 5
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 2
Blood pressure decreased (Investigations) | 0 | 3
Blood urine present (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 6
Lymphocyte count decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Respiratory rate increased (Investigations) | 0 | 1
Transaminases (Investigations) | 0 | 2
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Dermal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 10
Insomnia (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 10
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 8
Skin Infiltration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic dilatation (Vascular disorders) | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes